CLINICAL TRIAL: NCT05232474
Title: Implementation and Evaluation of a Guideline-based Clinical Decision Support System (KomPas+) Used by Therapists and Patients in the Treatment of Intermittent Claudication: a Cluster Randomized Trial With a Parallel Process Evaluation
Brief Title: Using KomPas+ in the Treatment of Patients With Intermittent Claudication
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other); Chronisch ZorgNet (Unknown); Koninklijk Nederlands Genootschap voor Fysiotherapie (Unknown); Vereniging van Oefentherapeuten Cesar en Mensendieck (Unknown); Harteraad (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021-13373
Record Dates: First submitted 2022-01-18; First posted 2022-02-09 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2023-03

CONDITIONS: Intermittent Claudication; Peripheral Arterial Disease
MeSH Terms: conditions — Intermittent Claudication; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group: no access to KomPas+ (Other): Therapists in the control group will not have access to KomPas+ and will continue to deliver usual care by using the KNGF guideline. They will also maintain access to KomPas. As with KomPas+, therapists are free to choose whether to use KomPas or not. The use of KomPas will also be encouraged.
  Interventions: Device: KomPas
- Experimental group: access to KomPas+ (Experimental): KomPas+ will be implemented within the experimental group. The use of KomPas+ in the physiotherapeutic treatment of patients with intermittent claudication will not be mandatory but will be encouraged through an implementation strategy. Therapists are free to choose whether to use it or not.
  Interventions: Device: KomPas+; Device: KomPas

INTERVENTIONS:
Device: KomPas+ — KomPas+ is a guideline-based clinical decision support system. With KomPas+, the aim is to integrate KomPas with the guideline recommendations for the conservative treatment process of patients with intermittent claudication. KomPas+ is a web-based tool, aimed to facilitate person-centered and participatory healthcare. Therapists have access to a tool that will help, for example, to improve consistency between patient-specific goals and the treatment plan. Using KomPas+, therapists are encouraged to discuss choices in the treatment plan with the patient. It is expected that the included topics in KomPas+ will not be burdensome for both patients and therapists. Topics to discuss are, for example, Frequency, Intensity, Time and Type (FITT) for drawing up a training schedule. KomPas+ is meant to facilitate therapists and patients in the SDM process. It does not force patients to take part in the SDM process against their will.
  Arms: Experimental group: access to KomPas+
Device: KomPas — KomPas is an online tool showing personalized outcome forecasts. These forecasts have been developed using real-world data of patients with intermittent claudication for physiotherapists in daily practice. The forecasts visualize the estimated outcome of supervised exercise therapy (walking distance and quality of life), for an individual patient with intermittent claudication. The information provided is based on patients similar to the individual patient from a large database. The actual outcome data of these similar patients are used to create an individual forecast. KomPas plots the estimated therapy outcome in time, thereby making personalized outcome forecasts. The forecasts are not used to direct the choices of treatment, but to motivate the patient, monitor the treatment process and to set realistic goals.

SUMMARY:
Intermittent claudication is the most common symptom of peripheral arterial disease (PAD). The recommended therapy is supervised exercise therapy combined with lifestyle counselling, provided by a physiotherapist. Ideally, during the treatment process patients' values and preferences are incorporated with evidence-based knowledge; shared decision making (SDM). Evidence shows the use of SDM in daily practice is scarce. Therefore, personalized outcome forecasts which provide insight into an individual's personal prognosis (called KomPas) were implemented in 2020. Now, as a next step, KomPas is further developed into a guideline-based clinical decision support system. The result is called KomPas+, a tool which integrates the person-centered approach of KomPas with the guideline recommendations for the conservative treatment of people with intermittent claudication.The primary objective of this study is to evaluate the impact of implementing KomPas+ in the physiotherapeutic treatment of patients with intermittent claudication on functional walking distance and health-related quality of life. Secondary, the level of SDM and person-centeredness of physiotherapists using KomPas or KomPas+ will be assessed. Third, the implementation process will be evaluated.

ELIGIBILITY:
Inclusion Criteria Primary objective:

- All therapists affiliated with Chronisch Zorgnet and specialized in the treatment of people with intermittent claudication are eligible to participate. Besides, all patients referred to a Chronisch Zorgnet therapist with intermittent claudication specialty are eligible to participate.

Inclusion Criteria Secondary objective:

* Provides written informed consent (both therapist and patients)
* Therapists should have finished two KomPas (control group) or KomPas+ (experimental group) e-learnings
* Therapists should have applied KomPas (control group) or KomPas+ (experimental group) to at least one patient with intermittent claudication

Inclusion Criteria Third objective:

- All therapists affiliated with Chronisch Zorgnet and specialized in the treatment of people with intermittent claudication who are included in the experimental group are eligible to participate.

Exclusion Criteria:

* Not applicable due to the "real world" setting of the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2271 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in Functional walking distance (FWD) using a standardized treadmill test at 3 months, 6 months, 9 months and 12 months. | Change from baseline at 3 months and 6 months
  The treadmill test is based on the graded Gardner-Skinner protocol. FWD is defined as the distance at which the patient would prefer to stop walking in daily life.
Mean Change from Baseline in Health-Related Quality of Life using the Vascular Quality of Life Questionnaire-6 (VascuQol-6) at 3 months, 6 months, 9 months and 12 months. | Change from baseline at 3 months and 6 months
  The VascuQol-6 consists of six questions related to activities, symptom burden, pain, emotions and social consequences. The score ranges from 6 to 24, with a higher score representing a better quality of life.

SECONDARY OUTCOMES:
Level of Person-Centredness assessed by using a Patient-Administered Questionnaire at the initial consult with the patient with intermittent claudication in which treatment goals and treatment plan are discussed. | During the initial consult with the patient with intermittent claudication in which treatment goals and treatment plan are discussed. This moment varies between the date of inclusion to three weeks after the date of inclusion.
  The used questions are part of the 36-item patient-centered primary care (PCPC) instrument.This Dutch instrument is specifically developed to assess person centered care in primary care setting for patients with multimorbidity. The complete PCPC instrument consists of 36 items divided over eight domains which are based on the eight dimensions of person centered care identified by the Picker Institute. For this study, the seven questions which form the subdomain 'Patients' preferences' are used. For example, patients will be asked if they felt taken seriously, if their wishes and preferences were taken into account and if they were involved in decisions about their treatment. Each of the seven questions will be responded by a five-point scale ranging from 1 (totally disagree) to 5 (totally agree) resulting in a total score between 7 and 35.
Level of Shared Decision Making (SDM) assessed by scoring video-records of clinical consultations with the Observer Patient Involvement (OPTION) 5 scale at the initial consult with the patient in which treatment goals and treatment plan are discussed. | During the initial consult with the patient with intermittent claudication in which treatment goals and treatment plan are discussed. This moment varies between the date of inclusion to three weeks after the date of inclusion.
  The five items of the OPTION-5 are based on the five core dimensions of SDM: alternate options (item 1), forming a partnership (item 2), inform about options (item 3), eliciting preferences (item 4), and integrate preferences (item 5). Each item will be scored on a five-point Likert scale from 0 (no effort) to 4 (exemplary effort) to obtain objective data of the SDM process. Item scores will be summed so that the potential total score is between 0 and 20. The total score will be rescaled to lie between 0 and 100.

OTHER OUTCOMES:
Perceived barriers and facilitators to (not) use KomPas+ in the physiotherapeutic treatment of patients with intermittent claudication using a qualitative assessment. | Between six and twelve months after the start of the implementation of KomPas+
  Semi-structured interviews within the experimental group. Both therapists who did use and did not use KomPas+ will be interviewed. The purpose will be to gain insight into why therapists did (not) use KomPas+, and therefore uncover ways to improve the uptake of using KomPas+ in the treatment of patients with intermittent claudication.
The degree of implementation of KomPas+ in terms of reach and demand measured by website logs (demand) and the use of KomPas+ (reach). | After the 4-month inclusion period
  Within the experimental group, website logs will show how many therapists completed multiple e-learnings aimed at (learning to use) KomPas+ (demand). Besides, it will be measured for how many newly referred patients KomPas+ is used during the inclusion period of the study, versus the number of new patients for which KomPas+ was not used. The difference gives an indication of the scope of the implementation (reach).

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Hoogeboom, PhD, Principal Investigator — Radboud university medical center, IQ healthcare
Locations (1):
- IQ healthcare, Radboudumc, Nijmegen, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data sets for publications related to the topic of this study will be published under restricted access. Publications will be made visible through the Radboud Repository including metadata describing the properties of the data. To access the data, a request needs to be submitted.